CLINICAL TRIAL: NCT04860414
Title: Prospective Monocentric Study of Taste in Patients With Minor or Major Cognitive Disorders Such as Alzheimer's, Through the Analysis of Gustatory Evoked Potentials
Acronym: MAPEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JACQUIN 2020
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Blood Specimen Collection; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Major Cognitive Impairment (Experimental)
  Interventions: Biological: Blood sampling; Other: Cognitive Assessment; Other: Subjective taste tests; Other: Objective taste tests
- Minor Cognitive Impairment (Experimental)
  Interventions: Biological: Blood sampling; Other: Cognitive Assessment; Other: Subjective taste tests; Other: Objective taste tests
- No Cognitive Impairment (Active Comparator)
  Interventions: Biological: Blood sampling; Other: Cognitive Assessment; Other: Subjective taste tests; Other: Objective taste tests

INTERVENTIONS:
Biological: Blood sampling — Fasting blood glucose, dosage of acylated and non-acylated ghrelin, leptin, insulin and serotonin.
Other: Cognitive Assessment — QPC Cognitive complaint questionnaire, CDR functional autonomy scales and IADL 4 items, MMSE cognitive scores, Dubois 5-word test, clock test, BREF, Isaacs test, BARD naming battery and MADRS depression scale
Other: Subjective taste tests — Scales of taste perceptive intensity, taste pleasure, hunger sensation (visual analogue scales from 0 to 10 cm) and food preferences on the one hand, and on the other hand, subjective tests of taste threshold determination by triangular tests of increasing sugar solution concentrations.
Other: Objective taste tests — Recording of gustatory evoked potentials

SUMMARY:
Approximately 24 million people worldwide suffer from dementia, with Alzheimer's disease being the most common cause. Alzheimer's disease typically progresses in three stages: presymptomatic, prodromal ("early onset" or minor cognitive impairment) and major cognitive impairment with loss of autonomy and significant psycho-behavioral symptoms. Efforts to counteract its expansion are increasing, and there is a need for biomarkers to identify the disease in its earliest stage in order to provide prompt treatment.

Faced with a episodic memory disorder, it is possible, thanks to certain criteria, highlighted by neuroimaging, or by biomarkers obtained by biological analysis of cerebrospinal fluid (during a lumbar puncture), to detect Alzheimer's disease from the prodromal stage, or even earlier. The main limitation of these criteria is their invasive nature. Other non-invasive biomarkers would therefore be useful to help diagnose Alzheimer's disease at an early stage. Gustatory evoked potentials (GEP), a technique for exploring taste sensory pathways, could meet these needs.

Indeed, GEPs are a method of exploring the gustatory sensory pathway based on the recording of cerebral electrical activity by electroencephalography (EEG). It is a painless, accessible, inexpensive and non-invasive technique. The alteration of gustatory functions is present in many neurological conditions, but often takes second place to sensory or motor symptoms. Rare studies have studied taste in patients with Alzheimer's disease, but they have demonstrated, using subjective tests only, an early gustatory impairment linked to a degeneration of the gustatory cortex. It was observed that the performance of subjects with minor or major cognitive impairment was weaker than that of healthy subjects, without the patient being aware of these taste disorders.

The aim of the study is to explore taste functions in patients with minor cognitive impairment, major cognitive impairment such as mild Alzheimer's disease, by comparing them to healthy subjects. For this purpose, we wish to compare the results of subjective taste tests (tasting solutions, especially salty ones, answering food preference questionnaires), parameters of taste evoked potentials recorded by electrodes stuck on the scalp and hormonal parameters obtained by blood sampling, between the three groups of subjects mentioned.

ELIGIBILITY:
Inclusion Criteria:

* A person who has given oral consent.
* For patients with early stage Alzheimer's disease, both the primary caregiver and the patient will need to give oral consent.
* ADULT
* Body Mass Index (BMI) < 30 kg/m².
* Patients meeting the diagnostic criteria for early-stage Alzheimer's disease: imaging (cerebral MRI), neuropsychobiological criteria (consultation with neuropsychological assessment, CSF biomarkers) and CDR (Clinical Dementia Rating Scale) rated at 1 or 1.5 - for the "subjects with early-stage Alzheimer's disease" group
* Patients meeting the diagnostic criteria for minor cognitive impairment: imaging (brain MRI) and neuropsychological assessment with a CDR scale of 0.5 - for the group "subjects with minor cognitive impairment".
* Absence of cognitive problems and normal neurological assessment - for the healthy group.
* Fasting at least 2 hours before PEG measurement

Exclusion Criteria:

* - A person who is not affiliated to or not a beneficiary of a social security system.
* Person subject to a measure of legal protection (curatorship, guardianship)
* Person subject to a judicial safeguard measure
* Pregnant, parturient or breastfeeding woman
* Adult unable to express consent or perform cognitive testing.
* Minor
* No Caregiver for Mild Alzheimer's Disease Patients
* Active smoker
* Diabetes (type 1 or type 2)
* Taking a treatment that interferes with taste
* Body Mass Index (BMI) ≥ 30 kg/m2
* MMS Score <20
* Cerebral MRI finding another cause of neurocognitive disorder (except for Fazekas 1 vascular lesions accepted).
* Known COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Amplitude of gustatory evoked potentials | After a fasting period of 2 hours
Latency of the gustatory evoked potential | After a fasting period of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] El Kadiri W, Perrignon-Sommet M, Delpont B, Graber M, Mohr S, Mouillot T, Devilliers H, Grall S, Lienard F, Georges M, Brindisi MC, Brondel L, Bejot Y, Leloup C, Jacquin-Piques A. Changes in Taste Perception in Patients with Minor and Major Cognitive Impairment Linked to Alzheimer's Disease Recorded by Gustatory Evoked Potentials. J Alzheimers Dis. 2023;96(4):1593-1607. doi: 10.3233/JAD-230270. PMID 38007646